CLINICAL TRIAL: NCT05173610
Title: Stereotactic Ablative Radiotherapy for Oligometastatic Hepatocellular Carcinoma: Phase II Trial
Brief Title: Stereotactic Ablative Radiotherapy for Oligometastatic Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1101
Record Dates: First submitted 2021-11-23; First posted 2021-12-30 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Oligometastasis Hepatocellular Carcinoma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT arm (Experimental): Patients will be treated with stereotactic body radiotherapy (SBRT) for oligometastasis from hepatocellular carcinoma
  Interventions: Radiation: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Radiation: Stereotactic body radiotherapy (SBRT) — Patients will be treated with stereotactic body radiotherapy (SBRT) for oligometastasis from hepatocellular carcinoma.
  1. Target delineation The GTV is set using diagnostic CT, MRI, PET-CT, etc. CTV is delineated including the microscopic range in GTV and internal margin using 4D-CT. The PTV is expanded by considering the uncertainty of the daily patient posture setting and placement.
  2. Radiotherapy All patients are treated using 3D-CRT, IMRT, or VMAT. Total dose and fractionations will be determined depending on the location and character of the metastasized tumor. Detailed radiation prescriptions is summarized in the following paragraph.
     i. Liver: 48-60 Gy in 4 fractions ii. Lung: 45-60 Gy in 3-4 fractions iii. Brain: 27-30 Gy in 3-5 fractions iv. bone: 24-40 Gy in 3-5 fractions v. adrenal gland: 30-60 Gy in 3-8 fractions vi. other organ: depending on the clinicians' decision

SUMMARY:
Oligometastasis is a definition that has been described in the past in the 1990s, and in some patients, metastases are not extensive and are limited to a small number of metastases. The local ablative treatment for oligometastasis is not a new concept. In case of liver metastasis from colorectal cancer, long-term survival can be expected if the liver resection is performed. Effectiveness has been demonstrated in studies of adrenal and brain metastasis from lung cancer as well as lung metastasis from sarcoma. A recent non-randomized study reported that patients with oligometastasis improved treatment outcomes with aggressive treatment. This study demonstrated that local ablative treatment for oligometastasis showed better treatment outcomes than expected. Also, the long-term outcomes in SABR-COMET trial showed that the overall survival were increased by 22 months. So far, the standard treatment for metastatic disease is systemic chemotherapy. However, based on these results from studies, active local treatment for patients with oligometastasis is currently being performed in the clinic. In this study, we aimed to apply this concept to patients with hepatocellular carcinoma. To confirm the efficacy and safety of stereotactic radiotherapy in patients with oligometastasis hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

i. 19 years or older

ii. Patients who signed the informed consent form

iii. The clinical trial protocol can be complied with at the discretion of the investigator

iv. Performance status (based on ECOG) less than 2 (0, 1)

v. Patients with life expectancy greater than 3 months

vi. Condition in which primary cancer is controlled

• Definition: A condition that has not progressed at the time of review of clinical trials after curative treatment of primary cancer 3 months ago

vii. Number of metastatic lesions up to 5

viii. 3 or less metastatic lesions in one metastatic organ

ix. Those who are undergoing targeted therapy or chemotherapy can also be included (during radiation therapy, drug treatment is stopped)

Exclusion Criteria:

i. Serious medical complications that cannot proceed with radiation therapy

ii. Previous radiation therapy history at the location where radiation therapy is to be performed

iii. malignant pleural effusion

iv. When the spinal cord and the tumor are close (the tumor is located within 3 mm)

v. In case of brain metastasis requiring surgical intervention

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-27 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy (Overall survival) | 2 year
  The overall survival of patients from the start date of SBRT to either date of death or date of last follow up is evaluated
Treatment efficacy (Disease free survival) | 2 year
  The disease free survival from the start date of SBRT to date of disease progression or date of death or date of last follow up is evaluated

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (acute and late toxicity) as assessed by CTCAE v4.0 | 2 year
  The acute and late treatment-related toxicity are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsil Seong, Principal Investigator — Department of radiation oncology, Yonsei cancer center, Yonsei University College of Medicine,
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
In case that individual participant data is being shared, the study protocol is planned to be shared.

REFERENCES:
- [Derived] Choi SH, Lee BM, Kim J, Kim DY, Seong J. Efficacy of stereotactic ablative radiotherapy in patients with oligometastatic hepatocellular carcinoma: A phase II study. J Hepatol. 2024 Jul;81(1):84-92. doi: 10.1016/j.jhep.2024.03.003. Epub 2024 Mar 11. PMID 38467379